CLINICAL TRIAL: NCT04366557
Title: The Influence of the Body Posture Correcting Therapy on Pelvic Floor Muscles Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katarzyna Jórasz (Other)
Responsible Party: Sponsor-Investigator, Katarzyna Jórasz, Principal Investigator, Józef Piłsudski University of Physical Education
Organization: Józef Piłsudski University of Physical Education (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKE 01-32/2018
Record Dates: First submitted 2020-04-18; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Musculoskeletal Manipulations; Exercise; Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Participants divided into two groups (the study and the control)
Who Masked: Participant
Masking Description: Subjects covered by the assigned number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body posture correction (Experimental): Subjects from study group had an education about pelvic floor and additional a six week body posture therapy.
  Interventions: Other: Manual therapy, exercises and education program
- Without correction of body posture (Other): Subjects form control group had only an education about pelvic floor.
  Interventions: Other: Education program

INTERVENTIONS:
Other: Manual therapy, exercises and education program — a six week body posture therapy consisted of manual therapy (once per week) and home exercises; education about pelvic floor
  Arms: Body posture correction
Other: Education program — education about pelvic floor
  Arms: Without correction of body posture

SUMMARY:
The purpose of this study is to assess the influence of the body posture correcting therapy on pelvic floor muscles function and urinary incontinence problem.

DETAILED DESCRIPTION:
This randomized, controlled study was aimed to asses influence of a six week global posture correction therapy on pelvic floor muscles function and urinary incontinence problem. Participants were randomly divided into two groups. All subjects overcame assessment of pelvic floor muscles (sEMG, manometry and digital) and completed questionnaire about urinary incontinence problem and general health condition connected with lower tract symptoms. Both groups had a pelvic floor education (what is it, where are the pelvic floor muscle, how to correct contract them etc.) Additionally, the study group had a six week therapy focused on body posture correction. Therapy consisted of manual therapy (once per week) and correction exercises.

ELIGIBILITY:
Inclusion Criteria:

* stress urinary incontinence (confirmed by a medical examination)
* female
* age between 25 and 45 years old

Exclusion Criteria:

* gynecological, spinal, and abdominal surgery (excluding cesarean delivery)
* menopause
* spinal and pelvis injuries
* chronic diseases of the circulatory and respiratory system
* neurlogical accidance

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF) | 6 week (post-treatment)
  evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence; scoring scale 0-21 (higher scores mean a worse outcome)
Change in Oswestry Disability Index (ODI) | 6 week (post-treatment)
  level of disability connected with chronic lumbar pain; scoring scale 0-50 (higher scores mean a worse outcome)
Change in King's Health Questionnaire (KHQ) | 6 week (post-treatment)
  to assess the impact of lower urinary tract symptoms including urinary incontinence on health related quality of life; the questionnarie consists of three parts; scoring scale: I-II part 0-100; III part 0-30 (higher scores mean a worse outcome)
Change in sEMG of the pelvic floor muscles | 6 week (post-treatment)
  using vaginal probe; average maximum voluntary isometric contraction and relaxation (after 5 attempts); unit of measure - mV (microvolts); higher scores mean a better outcome (contraction); higher scores mean the worse outcome (relaxation)
Change in manometry of the pelvic floor muscles | 6 week (post-treatment)
  to assess the pressure levels performed by voluntary contraction of pelvic floor muscles (after 5 attempts); unit of measure - centimeter of water column (cmH2O); higher scores mean the better outcome
Change in digital palpation of the pelvic floor muscles using PERFECT shame | 6 week (post-treatment)
  to assess power of pelvic floor muscles (P) - scoring scale 1-5 (higher is better), endurance (E) - scoring scale (higher is better), the ability to repeat the contraction with maximum strength (R) - scale 1-10 (higer is better); number of fast contractions (F) - scale 1-15 (higher is better); possibility of elevation of perineum (E) - yes/no; co-contraction of another muscles (C) - yes/no; involuntary contraction during coughing (T) - yes/no

CONTACTS AND LOCATIONS:
Locations (1):
- The rehabilitation clinic PROFEMED, Warsaw, Poland